CLINICAL TRIAL: NCT01913002
Title: Randomized, Double-blind, Placebo-controlled, Positive-controlled, 4-period, 4-way Crossover Study to Define the Electrocardiogram Effects of a Single Dose of LX4211 800 mg and 2000 mg Compared With Placebo and Open-label Moxifloxacin in Healthy Subjects: A Thorough QT Study
Brief Title: Study to Define the Electrocardiogram Effects of a Single Dose of LX4211 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LX4211.1-109-NRM; LX4211.109 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
MeSH Terms: interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): LX4211 800 mg
  Interventions: Drug: LX4211 800 mg; Drug: LX4211 2000 mg; Drug: moxifloxacin 400 mg; Drug: LX4211 Placebo
- Treatment B (Experimental): LX4211 2000 mg
  Interventions: Drug: LX4211 800 mg; Drug: LX4211 2000 mg; Drug: moxifloxacin 400 mg; Drug: LX4211 Placebo
- Treatment C (Active Comparator): moxifloxacin 400 mg
  Interventions: Drug: LX4211 800 mg; Drug: LX4211 2000 mg; Drug: moxifloxacin 400 mg; Drug: LX4211 Placebo
- Treatment D (Placebo Comparator): Placebo
  Interventions: Drug: LX4211 800 mg; Drug: LX4211 2000 mg; Drug: moxifloxacin 400 mg; Drug: LX4211 Placebo

INTERVENTIONS:
Drug: LX4211 800 mg
Drug: LX4211 2000 mg
Drug: moxifloxacin 400 mg
Drug: LX4211 Placebo

SUMMARY:
This Phase 1 study is to investigate the effects of higher doses of LX4211 (800 mg and 2000 mg) do not differ from placebo in the mean change in QTcI from Baseline in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects ≥18 to ≤55 years of age
* Vital signs at Screening in the following ranges: systolic blood pressure, 90-140 mmHg; diastolic blood pressure, 50-90 mmHg; heart rate, 45-100 bpm
* Body mass index (BMI) ≥18 and ≤35 kg/sq m
* Able and willing to provide written informed consent
* Nonsmoker and has not used any tobacco products for at least 3 months prior to Screening
* Willing to adhere to the prohibitions and restrictions specified in this protocol
* Able to tolerate prolonged periods of quiet, motionless, supervised rest

Exclusion Criteria:

* Use of any medication (prescription, over-the-counter, herbal tea, or supplements) within 5 days of dosing
* Use of any investigational agent or study treatment within 30 days prior to Screening
* Use of any protein or antibody-based therapeutic agents within 3 months prior to Screening
* Prior exposure to LX4211
* Daily use of cigarettes or any tobacco products within 3 months prior to Screening and while participating in the study
* History of any major surgery within 6 months prior to Screening
* History of any serious adverse reaction or hypersensitivity to any inactive component of LX4211
* History of renal disease or significantly abnormal kidney function tests
* History of hepatic disease or significantly abnormal liver function tests
* Women who are breastfeeding or are planning to become pregnant during the study
* History of any active infection within 14 days prior to Screening
* History of alcohol or substance abuse within 2 years prior to Screening
* History of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), HIV-1 or HIV-2
* Presence of clinically significant physical, laboratory, or ECG findings (eg, QTcF >450 msec for females and QTcF >430 msec for males) at Screening
* >30 premature ventricular beats per hour on the telemetry ECG monitoring at Day -2 of Period 1
* History of additional risk factors for the presence of a family history of Short QT Syndrome, Long QT Syndrome, sudden unexplained death at a young age (<=40 years), drowning or sudden infant death syndrome in a first degree relative (ie, biological parent, sibling, or child)
* Any skin condition likely to interfere with ECG electrode placement or adhesion
* Any skin condition likely to interfere with ECG electrode placement or adhesion
* Donation or loss of >400 mL of blood or blood product within 3 months prior to Screening
* Positive urine glucose during Screening
* Positive pregnancy test during Screening
* Positive urine screen for drugs of abuse during Screening
* Positive urine test for alcohol during Screening
* Inability or difficulty swallowing whole tablets or capsules
* Unable or unwilling to communicate or cooperate with the Investigator for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTc intervals | Day -1, Day 1 of each period (2, 3, 4)

SECONDARY OUTCOMES:
Number of subjects experiencing an adverse event | up to 87 days
Plasma concentrations of LX4211 | Day 1 of each Period: predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48, and 60 hours after dosing time on Day 1 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ikenna (Ike) Ogbaa, M.D., Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, Austin, Texas, United States